CLINICAL TRIAL: NCT04998227
Title: Latent TGF-β-binding Proteins Affect the Fibrotic Process in Renal Impairment and Cardiac Dysfunction
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202103008RINB
Record Dates: First submitted 2021-08-03; First posted 2021-08-10 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Acute Coronary Syndrome; Acute Coronary Syndrome With Renal Dysfunction
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- suspect acute coronary syndrome: Subjects with the diagnosis of suspected acute coronary syndrome (ACS), age between 20 to 80.
  Exclusion criteria: pregnant women, patients with end-stage renal disease (eGFR <15 mL/min/1.73 m2), cardiogenic shock.

SUMMARY:
The project is planed to explore the impact of LTBP4 and other matrix protein and potentially related biomarkers on renal outcomes, cardiac outcomes and all-cause mortality in patients with suspected acute coronary syndrome (ACS).

DETAILED DESCRIPTION:
The investigators will collect the blood samples from patients with suspect ACS. LTBP4 will be the first matrix protein that are going to understand. Upon hospital arrival, blood samples around 8 ml will be collected and the 2nd collection will be two weeks to one month after the event. The third collection will be one year later. In the between, if any ACS event develop, blood samples will be collected as protocols.

ELIGIBILITY:
Inclusion Criteria:

- acute coronary syndrome patients

Exclusion Criteria:

- cardiogenic shock, pregnancy, end-stage renal disease

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects between 20-80 yrs, with acute coronary syndrome in NTUH.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-04-26 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Change of renal functions | One month, Six month and one year
  The investigators will follow up Cr and eGFR levels correlate with LTBP4 levels
All cause mortality | 3 years
Incidence of hospitalization | 3 years
Incidence of required myocardial revascularization | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided